CLINICAL TRIAL: NCT01815008
Title: PHARMACOGENOMICS OF ANTI-PLATELET RESPONSE - I
Brief Title: Pharmacogenomics of Antiplatelet Response - I
Acronym: PARes-I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rehan Qayyum, Assistant Professor of Medicine, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: K23HL105897-PARes-I; K23HL105897 (NIH)
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Platelet Aggregation; Platelet Transcriptome; Coronary Artery Disease
Keywords: Platelet aggregation; Clopidogrel; Platelet transcriptome
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clopidogrel (Experimental): Clopidogrel 75 mg daily by mouth for 1 week then Clopidogrel 75 mg daily with aspirin 81 mg daily
  Interventions: Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75 mg daily
  Other Names: Plavix
Drug: Aspirin — Aspirin 81 mg daily

SUMMARY:
This clinical trial is examining the role of genetic polymorphism on the effect of clopidogrel (with or without aspirin) on platelet response in persons at high-risk for myocardial infarction or stroke due to family history of early-onset coronary artery disease.

DETAILED DESCRIPTION:
The main goal of this study is to explore the impact of the PEAR1 genetic variant (rs12041331) on responsiveness to clopidogrel. The investigators will further assess the role of other genetic variants in determining the response to single or dual anti-platelet therapy. Apparently healthy subjects (N= 2108) from high-risk families are being (a) identified from a proband with early-onset CAD and (b) genotyped on the Illumina 1 million platform, with imputation to 2.5 million single nucleotide polymorphisms. The investigators plan to characterize the variance in platelet aggregation to multiple agonists (ADP, collagen, and arachidonic acid) after 1-week therapy with clopidogrel in a high-risk subset of GeneSTAR subjects (N=100). The investigators further plan to determine the extent to which variants identified in the PEAR1 gene modify platelet responsiveness to inhibition by clopidogrel in this high-risk subset. In addition, the investigators aim is to determine the extent to which variants in other recently discovered genes, by themselves, and in combination with PEAR1, modify platelet responsiveness to clopidogrel alone and with aspirin in this high-risk subset. Lastly, the investigators also want to determine what changes in platelet mRNA are produced by aspirin alone and by aspirin with clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Participants from the GeneSTAR cohort
* Unaffected with no overt coronary artery disease or serious vascular event (stroke or peripheral vascular disease diagnosis
* Presence of an occult coronary artery disease phenotype as defined by coronary artery calcium scores about the MESA (Multiethnic Study of Atherosclerosis) 75th percentile for age sex, and race or ≥ 1 stenoses in any of the major coronary arteries or main branches of > 50%, or coronary plaque volumetric scores above our own 75th percentile, or any combination on cardiac computed tomographic angiography (performed recently as part of the GeneSTAR study and present for all persons being recruited)/
* Presence of occult cerebrovascular disease defined as presence of white matter hyperintensities (WMH) thought to represent ischemic small vessel cerebrovascular disease, and /or the presence of lacunes (old small strokes), or the presence of an Atherosclerosis Risk in Communities Study (ARIC) silent stroke score on a visual analogue scales of 4 or more (on a scale of 0-9).
* Women who are postmenopausal.
* Women who use a reliable contraceptive method; a reliable contraceptive method will be defined as personal history of tubal ligation, ongoing use of intra-uterine device, or ongoing use of oral contraceptive pills.

Exclusion Criteria:

* Presence of any CAD or stroke, transient ischemic attacks, peripheral arterial disease
* Persons taking aspirin, NSAIDS, or any anti-coagulants who are medically unable to stop them for a two week pre-trial
* A history of allergy to aspirin or clopidogrel
* Weight < 60kg
* Age < 45 and > 75 years of age
* A history of recent or any active bleeding
* Serious or current co-morbidity (AIDS, cancer)
* Pregnant women as determined by urine dipstick pregnancy test
* Any aneurysms on cranial magnetic resonance imaging/magnetic resonance angiography (obtained recently in the GeneSTAR participants)
* Blood pressure above >=159/95mmHg
* History of a gastric or duodenal ulcer, or significant gastrointestinal disease, like regional enteritis
* Mental incompetence to make a decision to participate (developmentally disabled, and persons with diagnosed psychiatric disorders-documented in primary care records).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rehan Qayyum, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- See also: GeneSTAR Research Program — http://www.genestarstudy.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clopidogrel
Started | 19 (Had difficulty in completing enrollment)
Completed | 15 (transcriptomic data was available on 9 participants only)
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Clopidogrel
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (5.2)
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race/Ethnicity, Customized [Number; unit: participants]
  African Americans | 14

OUTCOME MEASURES:

1. Primary Outcome: Difference in ADP-induced Platelet Aggregation
Description: ADP-induced platelet aggregation will be measured using impedance aggregometry in whole blood before and after 1-week of clopidogrel. The difference between the baseline and after clopidogrel therapy will be determined. Higher impedance represent higher platelet aggregation.
Time Frame: at baseline and at 1 week
Population: Data was collected before and after one week of clopidogrel. We found it difficult to enroll patients with low risk to the combined aspirin and clopidogrel and hence study was continued for the first week only.
Measure: Mean (Standard Deviation); unit: Difference in ohms (Post-Pre)
Arm/Group | Clopidogrel
Number analyzed (Participants) | 14
Difference in ohms (Post-Pre) | -5.2 (4.1)

2. Secondary Outcome: Difference in Arachidonic Acid-induced Platelet Aggregation
Description: Arachidonic Acid-induced platelet aggregation will be measured using impedance aggregometry in whole blood before and after 1-week of clopidogrel. The difference between the baseline and after clopidogrel therapy will be determined
Time Frame: At baseline and after 1-week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Difference in ohms (Post-Pre)
Groups:
- Clopidogrel: Clopidogrel 75 mg daily by mouth for 1 week then Clopidogrel 75 mg daily with aspirin 81 mg daily
  Clopidogrel: Clopidogrel 75 mg daily
  Note: The 2nd week of the study was not performed as we could not find low risk population in our cohort who could be given both anti-platelets without increased estimated risk of bleeding.
Arm/Group | Clopidogrel
Number analyzed (Participants) | 14
Difference in ohms (Post-Pre) | -5.2 (4.4)

3. Secondary Outcome: Difference in Collagen-induced Platelet Aggregation
Description: Collagen-induced platelet aggregation will be measured using impedance aggregometry in whole blood before and after 1-week of clopidogrel. The difference between the baseline and after clopidogrel therapy will be determined
Time Frame: At Baseline and at 1 week
Population: Note: The 2nd week of the study was not performed as we could not find low risk population in our cohort who could be given both anti-platelets without increased estimated risk of bleeding.
Measure: Mean (Standard Deviation); unit: Difference in ohms (Post-Pre)
Arm/Group | Clopidogrel
Number analyzed (Participants) | 15
Difference in ohms (Post-Pre) | -1.13 (4.1)

4. Secondary Outcome: Changes in Platelet Transcriptome With Clopidogrel
Description: Platelet transcriptome will be examined before and after 1 week of therapy with clopidogrel and differences will be determined
Time Frame: At baseline and at 1 week
Population: Note: The 2nd week of the study was not performed as we could not find low risk population in our cohort who could be given both anti-platelets without increased estimated risk of bleeding. Note that the top most gene (CNOT2) with the lowest p-value is being reported.
Measure: Mean (Standard Error); unit: FPKM
Groups:
- Clopidogrel: Clopidogrel 75 mg daily by mouth for 1 week then Clopidogrel 75 mg daily with aspirin 81 mg daily
  Clopidogrel: Clopidogrel 75 mg daily
  Aspirin: Aspirin 81 mg daily
  Note: The 2nd week of the study was not performed as we could not find low risk population in our cohort who could be given both anti-platelets without increased estimated risk of bleeding.
Arm/Group | Clopidogrel
Number analyzed (Participants) | 8
FPKM | 13.7 (3.55)

ADVERSE EVENTS:
Arm/Group | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No